CLINICAL TRIAL: NCT01115062
Title: Comparison of Lidocaine/Tetracaine Patch (SyneraTM), 4% Liposomal Lidocaine Cream (LMX-4) and Placebo for Pain Reduction During Venipuncture in Children
Brief Title: Comparison of Synera Patch Versus LMX-4 Cream Versus Placebo Patch for Pain Reduction During Venipuncture in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carol Morreale (Other)
Responsible Party: Sponsor-Investigator, Carol Morreale, Clinical Pharmacist Specialist, CAMC Health System
Organization: CAMC Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-10-2182
Record Dates: First submitted 2010-04-15; First posted 2010-05-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Pain; Venipuncture; Anesthetics, Local
Keywords: Pain; Children; Local anesthetics
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Synera Patch (Experimental): Synera Patch (lidocaine 70 mg/ tetracaine 70 mg)
  Interventions: Drug: Synera Patch
- LMX-4 Cream (Experimental): LMX-4 (liposomal lidocaine 4%) cream
  Interventions: Drug: LMX 4 Cream
- Placebo Patch (Placebo Comparator): Placebo Patch
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Synera Patch — Synera Patch (lidocaine 70 mg/ tetracaine 70 mg) will be applied for 30 minutes to the venipuncture site
  Other Names: Synera
  Arms: Synera Patch
Drug: LMX 4 Cream — LMX 4 (4% liposomal lidocaine) cream (2g) will be applied under Tegaderm for 30 minutes to the venipuncture site.
  Other Names: LMX-4
  Arms: LMX-4 Cream
Drug: Placebo Patch — A placebo patch with the same properties as the Synera patch but without lidocaine/tetracaine will be administered for 30 minutes to the venipuncture site.
  Other Names: Placebo
  Arms: Placebo Patch

SUMMARY:
The purpose of this study is to compare the effect of Synera patch versus LMX-4 cream and placebo on the level of pain, observed distress, difficulty of venipuncture and skin side effects in children undergoing intravenous blood draw in the emergency setting or the phlebotomy lab.

DETAILED DESCRIPTION:
This study will compare the effectiveness of a patch applied for 30 minutes (Synera-lidocaine 70 mg/tetracaine 70 mg) with the effectiveness of a cream (LMX-4- 4% liposomal lidocaine) and a placebo patch applied for the same length of time in reducing pain due to needle sticks in children. One hundred fifty children and adolescents 5-17 years old admitted to emergency department or presenting to the phlebotomy lab. will be randomly placed in each group. Children will rate their level of pain using the Faces Pain Scale-Revised (FPS-R) before the medication is applied, after the medication is removed and after the needle stick. Parents and research observer will fill out the Observed Behavioral Distress (OBD) score. The phlebotomist will rate how difficult it was to perform the needle sticks. Any skin reaction seen by the investigator after the cream or patch is removed will be noted and compared among the three groups.

Subjects will be monitored from the time of enrollment to 5 minutes post phlebotomy.The Time Frame for which data will be presented is one (1) year.

ELIGIBILITY:
Inclusion Criteria:

* Children requiring venipuncture for medical care
* The ability to demonstrate proper understanding of the Faces Pain Scale-Revised (FPS-R)
* Parents of enrolled children need to be present during the procedure and be willing to rate their child's pain

Exclusion Criteria:

* Damaged or inflamed skin at the designated application site
* Known sensitivity to components of Synera or LMX-4 (lidocaine, tetracaine, or local anesthetics of the amide or ester type, PABA derivatives)
* Contraindications to Synera or LMX-4 use (severe hepatic disease, history of drug-induced methemoglobinemia, taking Class 1 antiarrhythmics)
* Use of analgesics during the past 24 hours
* Teenage female participants who are pregnant or lactating
* If in the attending's judgment the patient cannot wait wait 30 minutes for a blood drawn. These conditions include but are not limited to: sepsis, trauma, surgical emergencies, severe dehydration.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Face Pain Scale-Revised (FPS-R) | Before the medication application, after the medication removal and after the venipuncture
  The child's understanding of the FPS-R will be pretested. Using the scale, the child will rate the level of pain experienced before the medication (patch, cream) application, after the medication removal and after the venipuncture.

SECONDARY OUTCOMES:
Observed Behavioral Distress Scale (OBDS) | Before, during and after venipuncture
  The parent, and a blinded research observer will complete the Observed Behavioral Distress Scale (OBDS) tool, which evaluates the observed patient distress at placement of the tourniquet (before venipuncture), at the needle insertion (during venipuncture), and at the placement of the adhesive bandage (after venipuncture).
Draize Scale for Adverse Skin Reactions | After removal of the patch or Tegaderm
  The investigator will record the skin reactions after removal of the patch (active or placebo) or the Tegaderm.
Venipuncture Difficulty | After venipuncture
  After completing the venipuncture the phlebotomist will rate the difficulty of this procedure.

CONTACTS AND LOCATIONS:
Overall Officials: James M. Turner, DO, Principal Investigator — Charleston Area Medical Center, Emergency Department
Locations (1):
- Women and Children Hospital, Charleston, West Virginia, United States